CLINICAL TRIAL: NCT05306002
Title: Effects of a Nutritional Intervention in DNA Damage of Patients With Hereditary Breast and Ovarian Cancer Syndrome
Brief Title: Nutritional Intervention and DNA Damage of Patients With HBOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Juan Antonio Pineda Juárez, Researcher - Research Coordination, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCONOV001
Record Dates: First submitted 2020-03-28; First posted 2022-03-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: HBOC Syndrome; DNA Damage; Nutrition Therapy
Keywords: HBOC Syndrome; DNA Damage; Nutrition Therapy
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antioxidant therapy (Other): The patient will get a nutritional personalized treatment with the following characteristics: hypocaloric diet, rich in micronutrients related with DNA reparation and polyphenols, with the next distribution: 45% carbohydrates, 30% lipids, 25% protein, <10% saturated fats, >10% unsaturated fats, based on the recommendations of the American Institute for Cancer Research (AICR).
  Interventions: Combination Product: Antioxidant therapy

INTERVENTIONS:
Combination Product: Antioxidant therapy — Antioxidant therapy based in the following dietary components: Zinc, Selenium, Magnesium, carotenoids, indole-3-carbinol, curcumin, epigalactocatechin, caffeine, resveratrol, lycopene, genistein, phytoestrogens

SUMMARY:
Breast and Ovarian Cancer Syndrome (HBOC) is characterized by mutations in tumor suppressor genes such as BRCA1 and BRCA2, which increase the carrier's risk of developing breast and ovarian cancer, especially before 40. In this pathology the DNA damage is increased because there is a state of chronic inflammation, plus the antineoplastic treatments and changes in body composition result in oxidative stress. The inductions of epigenetic changes by a nutritional intervention with an specific distribution of macronutrients, micronutrients and polyphenols, not only ensures an optimal nutritional status, but also shows a decrease in oxidative stress, and therefore in DNA damage. The aim of this study is to assess if the DNA damage in patients with HBOC decreases after the nutritional intervention.

DETAILED DESCRIPTION:
Breast and Ovarian Cancer Syndrome (HBOC) is a genetic disease characterized by mutations in tumor suppressor genes such as BRCA1 and BRCA2, elevation of Reactive Oxygen Species (ROS), inflammation and DNA damage; all this as a result of the pathology itself. Antineoplastic treatments and changes in body composition such as malnutrition, cachexia and obesity lead to an increase of the inflammatory state. The induction of epigenetic changes by a nutritional intervention suggests that an hypo caloric diet, complex carbohydrates, polyunsaturated fatty acids, some amino acids, and some vitamins, minerals and polyphenols as well, can reduce DNA damage because of the interaction between mechanisms related with DNA stability and reparation, cellular replication, induction of apoptosis, and antioxidant systems. Previous studies report that using polyphenols supplements can reduce de DNA damage, but when the administration is only through food there's no benefit at all. So the aim of this study is to assess if the use of different micronutrients and polyphenols in conjoint can make synergism and reduce de DNA damage without the need of supplements.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with HBOC according to the Mexican Consensus of Breast Cancer
* Patients over 18 years who voluntarily agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients with end-stage chronic kidney failure, heart failure, liver failure, rheumatoid arthritis, non-inherited AC or HIV.
* Patients who carry out a structured exercise plan (rehabilitation) at the time of inclusion in the study.
* Patients who carry out a structured eating plan (adherence to diet) or who are consuming a food supplement at the time of inclusion in the study.
* Patients with significant primary clinical disorders: hematological (hemoglobin <13 in men and <12 in women), renal (creatinine> 3), neurological (other than epilepsy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
DNA damage change | 12 weeks
  A blood sample will be taken to assess DNA damage (ELISA) by 8-hydroxy-2-deoxyguanosine (8-OHdG), a modified nitrogen base indicating oxidative damage to DNA, before and after nutritional intervention.

SECONDARY OUTCOMES:
Body composition change | 12 weeks
  A bioelectrical impedance analysis will be used to assess the body composition through the reactance and resistance values (both measured in Ohm), before and after nutritional intervention.
Muscular strength change | 12 weeks
  A hand grip dynamometer will be used to assess the muscular strength in kg, both before and after the nutritional intervention.
Dietary change: Energy | 12 weeks
  A 24-hour recalls will be performed to evaluate amount of energy (measured in kilocalories), before and after the nutritional intervention.
Dietary change: Macronutrients | 12 weeks
  A 24-hour recalls will be performed to evaluate amount of carbohydrate, protein and fat (all measured in percentage and grams), before and after the nutritional intervention.
Dietary change: Micronutrients | 12 weeks
  A 24-hour recalls will be performed to evaluate amount of vitamin E, calcium, zinc and magnesium (all measured in milligrams), before and after the nutritional intervention.
  A 24-hour recalls will be performed to evaluate amount of folate, vitamin A and D, selenium, lycopene, and flavones (all measured in micrograms), before and after the nutritional intervention.

CONTACTS AND LOCATIONS:
Overall Officials: María Fernanda Díaz Yáñez, BSc, Principal Investigator — CMN "20 de Noviembre"; Martha Fernanda Medero López, BSc, Principal Investigator — CMN "20 de Noviembre"; Juan Antonio Pineda Juárez, PhD, Study Director — CMN "20 de Noviembre"; Martha Orozco Quiyono, MSc, Study Chair — CMN "20 de Noviembre"; Mónica Escamilla Tilch, PhD, Study Chair — CMN "20 de Noviembre"
Locations (1):
- María Fernanda Díaz Yáñez, Mexico City, Benito Juárez, Mexico

IPD SHARING:
Plan to Share IPD: No
Will individual participant data be available (including data dictionaries)? No
  What data in particular will be shared? Not available
  What other documents will be available? Study Protocol, Statistical will be available? Analysis Plan, Informed Consent Form, Clinical Study Report

REFERENCES:
- [Background] Kowalska E, Narod SA, Huzarski T, Zajaczek S, Huzarska J, Gorski B, Lubinski J. Increased rates of chromosome breakage in BRCA1 carriers are normalized by oral selenium supplementation. Cancer Epidemiol Biomarkers Prev. 2005 May;14(5):1302-6. doi: 10.1158/1055-9965.EPI-03-0448. PMID 15894690
- [Background] Kasai H. Analysis of a form of oxidative DNA damage, 8-hydroxy-2'-deoxyguanosine, as a marker of cellular oxidative stress during carcinogenesis. Mutat Res. 1997 Dec;387(3):147-63. doi: 10.1016/s1383-5742(97)00035-5. PMID 9439711
- [Background] Gopalakrishnan S, Van Emburgh BO, Robertson KD. DNA methylation in development and human disease. Mutat Res. 2008 Dec 1;647(1-2):30-8. doi: 10.1016/j.mrfmmm.2008.08.006. Epub 2008 Aug 20. PMID 18778722
- [Background] Ferguson LR, Chen H, Collins AR, Connell M, Damia G, Dasgupta S, Malhotra M, Meeker AK, Amedei A, Amin A, Ashraf SS, Aquilano K, Azmi AS, Bhakta D, Bilsland A, Boosani CS, Chen S, Ciriolo MR, Fujii H, Guha G, Halicka D, Helferich WG, Keith WN, Mohammed SI, Niccolai E, Yang X, Honoki K, Parslow VR, Prakash S, Rezazadeh S, Shackelford RE, Sidransky D, Tran PT, Yang ES, Maxwell CA. Genomic instability in human cancer: Molecular insights and opportunities for therapeutic attack and prevention through diet and nutrition. Semin Cancer Biol. 2015 Dec;35 Suppl(Suppl):S5-S24. doi: 10.1016/j.semcancer.2015.03.005. Epub 2015 Apr 11. PMID 25869442
- [Background] Higdon JV, Delage B, Williams DE, Dashwood RH. Cruciferous vegetables and human cancer risk: epidemiologic evidence and mechanistic basis. Pharmacol Res. 2007 Mar;55(3):224-36. doi: 10.1016/j.phrs.2007.01.009. Epub 2007 Jan 25. PMID 17317210